CLINICAL TRIAL: NCT05340543
Title: Ex-vivo Examination of Excisions of Skin Tumors by Confocal Optical Coherence Tomography (LC-OCT) With Integrated Dermoscopy and Comparison With Histology (DERMOCTAV)
Acronym: DERMOCTAV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02609-48
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-01

CONDITIONS: Cutaneous Tumor; Optical Coherence Tomography; Basal Cell Carcinoma; Squamous Cell Carcinoma; Melanoma
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with basal cell carcinoma: - CBC: Presence of lobule of basal cells with "palisading" on the edges, stromal reaction and dilated horizontal vessels.
  Interventions: Procedure: Confocal optical coherence tomography - OCTAVE
- Patient with squamous cell carcinoma: - CSC: Proliferation of keratinocytes presenting cellular atypia, crossing the JDE (invasive CSC versus in situ), glomerular vessels
  Interventions: Procedure: Confocal optical coherence tomography - OCTAVE
- Patient with melanoma: Melanoma: Destructured dermal-epidermal junction (DEJ), presence of pagetoid cells, clusters of atypical melanocytes, dendritic cells
  Interventions: Procedure: Confocal optical coherence tomography - OCTAVE

INTERVENTIONS:
Procedure: Confocal optical coherence tomography - OCTAVE — An ex vivo examination of cutaneous resection with the OCTAV® prototype integrating the "dermoscope" function

SUMMARY:
This project aims to validate ex vivo the use of the OCTAV® prototype integrating the "dermoscope" function before an in vivo application, by comparing images obtained by the OCTAV® prototype integrating the "dermoscope" function with the histological sections of a skin tumor excision corresponding to them exactly, at the same level.

DETAILED DESCRIPTION:
There are mainly 3 types of skin cancer: melanoma, basal cell carcinoma and squamous cell carcinoma. The diagnosis of skin cancers is now based on anatomo-pathological evidence. However, given the progress made, imaging is a technique that now has a full role in the diagnosis of these pathologies. This is particularly the case of confocal optical coherence tomography (LC-OCT), which is a recent imaging technique that has proven itself in ophthalmology with the obtaining of precise images of the retina.

LC-OCT can be applied in dermatology according to the following principle: the low intensity laser beam delivered by the LC-OCT device interferes with the melanin, is reflected and makes it possible to instantly acquire a 3D cross-sectional image of the skin, with a resolution of the order of a micrometer. It is finally an "optical echography", the light allowing a tissue definition much higher than the ultrasonic waves. It is therefore possible to obtain sections of histological resolution, and to scan the entire area studied.

Based on this principle, DAMAE has created OCTAV®, a class 1 medical device intended to allow "an in-depth study of skin pathologies", which is currently being evaluated in vivo as part of a clinical trial ( OCTAV - NCT03731247).

The device evaluated in the OCTAV trial does not include the "dermoscope" function. However, coupled with an image capture and processing system, it would increase the magnification obtained from 10 times to 20 or 30 times, allowing precise targeting of the lesion. As a result, a new prototype of OCTAV® has been developed which integrates the "dermoscope" function.

In this context, this project aims to validate ex vivo the use of the OCTAV® prototype integrating the "dermoscope" function before an in vivo application, by comparing images obtained by the OCTAV® prototype integrating the "dermoscope" function with the histological sections of a skin tumor excision corresponding to them exactly, at the same level.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, at least 18 years old
* Patient with a skin lesion suspected of a cancerous pathology (basal cell carcinoma - BCC, squamous cell carcinoma - SCC and melanoma) and for whom surgery is planned at Antony Hospital
* Affiliated patient or beneficiary of a social security scheme
* Patient having signed the free and informed consent

Exclusion Criteria:

* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant or breastfeeding women
* Patient hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a skin lesion suspected of a cancerous pathology (basal cell carcinoma - BCC, squamous cell carcinoma - SCC and melanoma) and for whom surgery is planned at Antony Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-06-16 (Estimated); Study Completion 2022-06-16 (Estimated)

PRIMARY OUTCOMES:
Concordance RATE | 10 days
  Correlation between LC-OCT images on the first 500 microns of the skin and histological images of skin and tumor excision analysis.

CONTACTS AND LOCATIONS:
Overall Officials: DRE RAMSAYGDS, Study Chair — Ramsay Générale de Santé
Locations (1):
- Hôpital Privé d'Antony Antony, Antony, IDF, France